CLINICAL TRIAL: NCT06731933
Title: Impact of Collagen VII Gene Therapy on Squamous Cell Carcinoma Recurrence in Recessive Dystrophic Epidermolysis Bullosa Skin
Brief Title: Impact of COL7A1 Gene Therapy on SCC Recurrence in RDEB Skin
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Epidermolysis Bullosa Research Partnership (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-73906
Record Dates: First submitted 2024-12-11; First posted 2024-12-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Squamous Cell Carcinoma
Keywords: gene therapy
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment with BVEC (Active Comparator)
  Interventions: Drug: BVEC
- No treatment with BVEC (No Intervention)

INTERVENTIONS:
Drug: BVEC — The study drug will be administered by home nurse at Subjects home for the participants residing in US. No drug will be applied when at study site. The subjects enrolled in Bari, Italy will not be administered BVEC.
  Other Names: Beremagene Geperpavec
  Arms: Treatment with BVEC

SUMMARY:
The study objective is to see if BVEC induced C7 expression in Recessive Dystrophic Epidermolysis Bullosa (RDEB) skin following Squamous cell carcinoma (SCC) excision will normalize the invasive tumor microenvironment and reduce tumor recurrence.

Prevention of SCC's in the RDEB subjects will increase their life span.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of generalized Recessive dystrophic epidermolysis bullosa (RDEB) demonstrated by COL7A1 mutations
2. Presence of biopsy proven squamous cell carcinoma (SCC)
3. Ability to understand and the willingness to provide written informed consent.
4. US based participants are willing to use beremagene geperpavec (BVEC)
5. Subject is 18 years or older
6. participant willingness to use an effective method of contraception

Exclusion Criteria:

1. Inability to travel to site for study visit
2. Subject is pregnant
3. Subject has Metastatic SCC's or is on any current systemic treatment for SCC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of Squamous Cell Carcinoma | 2 years
  The outcome measure is recurrence rate of SCC following BVEC application at each SCC lesion

CONTACTS AND LOCATIONS:
Overall Officials: Peter Marinkovich, MD, Principal Investigator — Stanford University
Locations (2):
- Stanford University, Redwood City, California, United States
- Azienda Ospedliero-Universitaia, Bari, Italy